CLINICAL TRIAL: NCT04373850
Title: Reducing Readmission Rates by Providing a Comprehensive Transition Plan From Hospital to Home for Cardiac Surgery Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00097613
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Cardiac Surgery
Keywords: Reducing readmissions
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home visit group (Experimental): Will receive a home visit after discharge in addition to the standard discharge planning.
  Interventions: Behavioral: Home Visit
- Control group (No Intervention): Will receive only the standard discharge planning.

INTERVENTIONS:
Behavioral: Home Visit — Physical exam, medication dose titration
  Arms: Home visit group

SUMMARY:
Patients who undergo cardiac surgery will be screened by a team member with the risk score once the patient has been admitted to the Cardiovascular Progressive Care Unit (CVPCU) after surgery. Participants will be randomized to the intervention or the control group. Both groups will receive standard discharge planning. In addition, the intervention group will have a nurse practitioner (NP) who will be responsible to verify that each essential step of the discharge process has been completed and will visit the patient in patient's home after discharge to complete a physical, review medications, titrate medications as needed, prescribe any necessary treatments, and perform education. The primary outcome variable will be a decrease in the 30 day readmission rate comparing high risk patients at pre and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or greater who have had cardiac surgery procedures including coronary artery bypass surgery (CABG), valve replacement, aortic aneurysm repair, and combined CABG and valve procedures.

Exclusion Criteria:

* Patients who have undergone orthotopic heart transplantation, orthotopic lung transplantation, or orthotopic heart-lung transplantation
* Patients who have undergone ventricular assist device placement
* Patients who do not reside in Maryland
* Non English speaking patients
* Patients discharged to a facility.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
30-Day readmission rate | Up to 30 days post discharge
  Rate of readmissions within 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Owens, PhD, Principal Investigator — Johns Hopkins University